CLINICAL TRIAL: NCT04315987
Title: Exploratory Clinical Study to Assess the Efficacy of NestaCell® Mesenchymal Stem Cell to Treat Patients With Severe COVID-19 Pneumonia
Brief Title: NestaCell® Mesenchymal Stem Cell to Treat Patients With Severe COVID-19 Pneumonia
Acronym: HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Cellavita Pesquisa Científica Ltda (Other); Hospital Vera Cruz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1) to receive NestaCell (n=45) or Placebo (n=45).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NestaCell® (Experimental): A dose of 2x10^7 cells (20 million cells) will be administered IV on days 1, 3, 5 and 7 in all subjects.
  Interventions: Biological: NestaCell®
- Placebo (Placebo Comparator): Matching placebo will be administered IV on days 1, 3, 5 and 7 in all subjects.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NestaCell® — A dose of 2x10^7 cells (20 million cells) will be administered IV on days 1, 3, 5 and 7 in all subjects.
  Other Names: Mesenchymal Stem Cell
  Arms: NestaCell®
Biological: Placebo — Matching Placebo will be administered IV on days 1, 3, 5 and 7 in all subjects.
  Arms: Placebo

SUMMARY:
This is phase II study to assess the efficacy of NestaCell® (mesenchymal stem cell) to treat severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
The number of infections of COVID-19 worldwide has killed thousands and is continually rising. The novel coronavirus attacks the human body by attaching to the angiotensin-converting enzyme-2 (ACE2), a protective enzyme against lung damage. In addition, the cellular serine protease TMPRSS2 for HCoV-19 Spike protein priming is also essential for the host cell entry and spread. Coronaviruses can be deadly, in large part because they cause "cytokine storms." These storms result from imbalances between pro-inflammatory and anti-inflammatory proteins called cytokines, which can cause extreme inflammation and respiratory complications. Respiratory distress kills hundreds of thousands of people each year worldwide, and hundreds of clinical trials are testing drugs to treat it.

MSCs have been widely used in cell-based therapy, from basic research to clinical trials Safety and effectiveness have been clearly documented in many clinical trials, especially in the immune-mediated inflammatory diseases.

NestaCell® is a mesenchymal stem cell therapy produced by Cellavita and proved to be safe in previous clinical trials.

The aim of this study is assess the efficacy of NestCell® as an add-on therapy to standard treatment to treat patients with severe COVID-19 pneumonia. .

Patients included will be randomized to receive 2x10^7 cells (20 million cells) on days 1, 3, 5 and 7.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years 2. Present a confirmed or pending diagnosis of COVID-19, but with tomographic and clinical signs strongly suggestive of SARS-CoV-2 infection (COVID-19), with pulmonary impairment greater than or equal to 50% and: i. Oxygen saturation <95%; ii. CURB-65 rating ≥ a 4; d) Participants with a score on WHO ordinal scale that measures illness severity over time equal to 5 (Hospitalized with non-invasive ventilation or high-flow oxygen).

Exclusion Criteria:

1. Patients with autoimmune diseases in the past or screening;
2. Those who have serious basic diseases that affect their survival, including: malignant tumor, hematopathy, malignant fluid, active hemorrhage, severe malnutrition, etc. which have not been controlled and can not be removed due to multiple metastasis;
3. Known or self-reported HIV or syphilis infected persons;
4. Have participated in stem cell clinical research;
5. Pregnant or lactating women or those who have fertility plans in the past year;
6. The estimated life cycle is less than 48 hours;
7. Other conditions that the researcher thinks are not suitable for participating in the experiment.
8. Shock
9. Continuous use of immunosuppressive agents or organ transplants in the past 6 months;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Condition | 10 days
  Ordinal scale (WHO ordinal scale that measures illness severity over time)

SECONDARY OUTCOMES:
Rate of mortality within 10-days | 10 days
  Evaluation of Pneumonia change
Change of Clinical symptoms - respiratory rate | 10 days
  Evaluation of Pneumonia change
Hypoxia | 10 days
  oxygen saturation
PaO2 / FiO2 ratio | 10 days
  oxygen saturation
CD4+ and CD8+ T cell count | Days 1, 2, 4, 6 and 8.
  Marker of Immunological function
Changes of blood oxygen | 10 days
  PaO2 / FiO2 ratio
Side effects in the treatment group | 10 days
  Number of participants with treatment-related adverse events
Complete blood count, cardiac, hepatic and renal profiles; | Days 1, 2, 4, 6 and 8.
  Complete blood count, ALT, AST, GGT, CK, CKmB and creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Florentino de Araujo Cardoso Filho, Principal Investigator — Hospital Vera Cruz
Locations (4):
- Brazil (4):
  - Hospital Vera Cruz, Campinas, São Paulo
  - Hospital de Barueri, São Paulo
  - IncCOR, São Paulo
  - UNIFESP, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data of the study will become public.